CLINICAL TRIAL: NCT06326658
Title: Evaluation of the Curative Effect and Health Economics of Bufei Yishen Prescription on Patients With Frequent Acute Exacerbation of COPD in Stable Stage
Brief Title: Bufei Yishen Prescription on Patients With Frequent AECOPD in Stable Stage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for Frequent AECOPD
Record Dates: First submitted 2024-03-08; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Bufei Yishen Prescription; AECOPD; remission period; frequent
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bufei Yishen Prescription (Experimental): Bufei Yishen formula consists of Radix Panax Ginseng 6g, Radix Astragali 15g, Cornu Cervi Pantotrichum 12g, Fructus Lycii 12g, Fructus Schisandrae Chinensis 9g, Fructus Epimedium Brevicornum 9g, Fructus Pelargonium Chinense 9g, Radix Paeoniae Lactiflorae 9g, Rhizoma Dillonis 9g, Fructus Ziziphiroxylon 9g, Fructus Schisandrae Chinense 15g, Pericarpium Citriodora 9g
  Interventions: Other: Bufei Yishen Prescription Granule
- Bufei Yishen Prescription placebo (Placebo Comparator): Bufei Yishen Prescription placebo is prepared by adding 5% of the drug on the basis of dextrin and bitter agent, and its appearance, weight, color and smell are consistent with Chinese medicine granules.
  Interventions: Other: Bufei Yishen Prescription Granule

INTERVENTIONS:
Other: Bufei Yishen Prescription Granule — The comparison group was given Bufei Yishen Prescription Granule.The course of treatment was the same as that of the experimental group.

SUMMARY:
To evaluate the clinical efficacy and health economic advantages of Lung Replenishing and Kidney Enhancing Formula for the treatment of patients with frequent acute exacerbations in the stabilized phase.

DETAILED DESCRIPTION:
This study is based on a real world using a multicenter, randomized, double-blind, placebo-controlled trial.Based on a real-world multi-center, randomized, double-blind, placebo-controlled trial, this study will clinically observe patients with frequent acute exacerbations of chronic obstructive pulmonary disease in the stable phase.The study will evaluate the clinical efficacy and safety of Chinese medicine treatment programs in patients with frequent acute exacerbations of stable chronic obstructive pulmonary disease, and provide high-quality evidence for the popularization and application of Chinese medicine therapy in chronic obstructive pulmonary disease.This study will scientifically evaluate the clinical efficacy and safety of TCM treatment programs in patients with frequent acute exacerbations of stable chronic obstructive pulmonary disease, and provide high-quality evidence for the popularization of TCM evidence-based treatment in chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COPD at a stable stage.
* Stable COPD patients with frequent acute exacerbation.
* Age 40-80 years old.
* The condition was stable 4 weeks before enrollment.
* 5 did not participate in other drug clinical studies within 1 month before enrollment.
* At least 3 months of maintenance therapy with triple inhalation preparation was used before enrollment.
* Washout period was 2 weeks before enrollment.
* Voluntarily receive treatment and sign informed consent.

Exclusion Criteria:

* complicity with other diagnosed and clinically significant respiratory diseases, including but not limited to: asthma, active pulmonary tuberculosis, bronchiectasis, pulmonary hypertension, pulmonary embolism, pneumothorax, pleural effusion, interstitial lung disease, or other active pulmonary diseases requiring intervention.
* Patients with severe or acute cardiovascular and cerebrovascular diseases (acute cardiovascular and cerebrovascular events, malignant arrhythmias, unstable angina pectoris, cardiac function grade 3 or above, uncontrolled hypertension, etc.).
* Complicated with severe liver and kidney disease (severe liver disease refers to cirrhosis, portal hypertension and varicose vein bleeding, serious kidney disease including dialysis, kidney transplantation).
* Any item of liver function index (ALT, AST) exceeds the upper limit of normal reference value by 1.5 times, and renal function index Scr exceeds the upper limit of normal reference value.
* Tumor patients who have undergone surgical resection, radiotherapy and chemotherapy in the past five years.
* Patients with mobility difficulties caused by severe osteoarthropathy, neuromuscular disease, and peripheral vascular disease.
* Combined with absolute or relative prohibition of 6-minute walking test: such as resting heart rate > 120 beats/min, systolic blood pressure > 180mmHg or diastolic blood pressure > 100mmHg; Or have limited activity to complete the 6-minute walking test.
* Combined with cognitive or mental disorders.
* Glucocorticoids were taken orally within 2 weeks before enrollment.
* Had taken any Chinese medicine preparations (decoction, formula granule, proprietary Chinese medicine, etc.) prohibited during the study period according to the protocol within 2 weeks before enrollment.
* People who are known to be allergic to therapeutic drugs.
* Pregnant and lactating women, people who plan to become pregnant or cannot use effective contraceptive measures.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The number of acute exacerbations | Change from baseline the number of acute exacerbations at month 3, 6, 9and 12.
  The number of acute exacerbations

SECONDARY OUTCOMES:
The number of AECOPD leading to hospitalization and death | Change from baseline the number of AECOPD leading to hospitalization and death at month 3, 6, 9 and 12.
  Deaths due to AECOPD should be recorded in the study diary.
Time of onset of the first AECOPD | Immediately after the intervention
  the interval between the first medication and the first AECOPD (days).
Severity of AECOPD | Change from baseline severity of AECOPD at month 3, 6, 9and 12.
  mild, moderate and severe
Duration of AECOPD | Change from baseline duration of AECOPD at month 3, 6, 9and 12.
  The duration of acute exacerbation is from the beginning of an acute exacerbation to the stabilization of the disease
Case fatality rate | Up to month 12
  including the case fatality rate of AECOPD and the all-cause case fatality rate
Lung function | Change from baseline lung function at month 3, 6, 9and 12.
  FVC, FEV1, FEV1 % of the estimated value, FEV1/FVC were mainly used for evaluation
Score for clinical signs and symptoms | Change from baseline clinical symptoms and signs at month 3, 6, 9and 12.
  Formulate with reference to the "Guidelines for Clinical Research of New Chinese Medicines"Clinical scoring is weighted or assigned according to some of the main symptoms, signs, physiological parameters of patients, etc., so as to quantitatively evaluate the severity of the disease.The higher the score, the worse the state.
6-minute walking distance (6MWD) | Change from baseline 6-minute walking distance (6MWD) at month 3, 6, 9and 12.
  The 6-minute walking test standard published by ERS and ATS was adopted
The Chronic Obstructive Pulmonary Patient Self-Assessment Test (CAT) | Change from baseline the chronic obstructive pulmonary patient self-assessment test (CAT) at month 3, 6, 9and 12.
  The Chronic Obstructive Pulmonary Patient Self-Assessment Test (CAT), with a score range of 0 to 40.The higher the score, the worse the state.
The MOS item short fromhealth survey（SF-36） | Change from baseline SF-36 scale at month 3, 6, 9and 12.
  SF-36 Includes 8 dimensions: physical functioning, physical functioning, somatic pain, general health status, social functioning, emotional functioning, and mental health.The higher the score, the worse the state.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao Q, Wang M, Li Z, Chen T, Li J. Efficacy and health economics of Bufei Yishen granules in patients with frequent exacerbator phenotype in the stable phase of chronic obstructive pulmonary disease: study protocol for a multicenter, randomized, double-blind, placebo-controlled trial. Front Med (Lausanne). 2025 Sep 3;12:1662655. doi: 10.3389/fmed.2025.1662655. eCollection 2025. PMID 40969810